CLINICAL TRIAL: NCT01718041
Title: A Long-acting Human Growth Hormone (VRS-317) in Pre-pubertal Children With Growth Hormone Deficiency: A Randomized, Open-label, Multi-center, Phase 1b/2a Study of Safety, Tolerability, Pharmacokinetics (PK), Pharmacodynamics (PD) and Efficacy After Subcutaneous Administration for 6 Months
Brief Title: Versartis Trial in Children to Assess Long-Acting Growth Hormone
Acronym: VERTICAL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Versartis Inc. (Industry)
Responsible Party: Sponsor
Organization: Aravive, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRS-317 Protocol 12VR2
Record Dates: First submitted 2012-10-19; First posted 2012-10-31 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Pediatric Growth Hormone Deficiency
Keywords: Growth hormone; Growth hormone deficiency; Growth; Pediatric growth hormone deficiency; Long acting growth hormone; GHD; PGHD; VRS 317; Exten; Versartis
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VRS-317 (Experimental): Active treatment arm
  Interventions: Drug: Experimental: VRS-317

INTERVENTIONS:
Drug: Experimental: VRS-317 — Active treatment arm

SUMMARY:
This is a Phase 1b/2a study of VRS-317 (long-acting growth hormone) in pediatric patients with growth hormone deficiency. During Phase 1b, pediatric patients each will receive a single subcutaneous injection of VRS-317. During the Phase 2a stage, patients will receive 6 months of VRS-317 treatment at dose levels selected from the Phase 1b stage. The primary endpoints for the study are to determine the safety and efficacy of repeat dose VRS-317.

DETAILED DESCRIPTION:
In Phase 1b, separate cohorts of patients will be tested in a single ascending dose format. Safety review committee meetings will take place prior to escalating to each increasing dose level. Enrolled patients will be monitored for 60 days for safety with PK/PD and safety labs collected.

Two dose levels will be selected after completion of Phase 1b to be tested during Phase 2a (6 months of continuous VRS-317 treatment). Safety and PK assessments will be made during the Phase 2a stage. Patient heights will be measured by stadiometer.

ELIGIBILITY:
Inclusion Criteria:

* Chronological Age ≥ 3.0 years and ≤ 11.0
* Diagnosis of GHD as documented by GH stimulation test
* Below average height SDS at screening
* Appropriate weight for Stature
* Decreased IGF-I SDS at screening
* Delayed bone age
* Normal thyroid function test results at screening visit
* Legally authorized representative informed consent.

Exclusion Criteria:

* Prior treatment with any growth promoting agent
* Documented history of, or current, significant disease
* Chromosomal aneuploidy, significant gene mutations
* Diagnosis of Attention Deficit Hyperactivity Disorder
* Daily use of anti-inflammatory doses of glucocorticoid
* Prior history of leukemia, lymphoma, sarcoma or cancer
* Known allergy to constituents of the study drug formulation
* Abnormal ocular findings at screening
* Significant abnormality in screening laboratory studies

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Phase 1b and 2a: Evaluate the safety and tolerability of multiple dosing levels of subcutaneous (SC) VRS-317 in pediatric growth hormone deficient (GHD) patients. Phase 2a: Evaluate the efficacy of multiple dose levels of VRS-317 | 8 Months
  Safety observations will include the number of patients with adverse events, concomitant medications, safety labs, vital signs, physical exams, single dose immunogenicity (Phase 1b), and repeat dose immunogenicity (Phase 2a).
  The primary efficacy outcome measure is the height velocity over 6 months as measured by standing height taken with stadiometer at baseline and after 6 Months of VRS-317 dosing in Phase 2a.

SECONDARY OUTCOMES:
Evaluate pharmacokinetic measures of VRS-317. | 8 months
  Secondary outcome measures include evaluation of pharmacokinetics (PK) of VRS-317 including Cmax, Tmax and AUC. PK measures will be analysed at multiple timepoints after single dosing of VRS-317 during Phase 1b and after repeat dosing of VRS-317 during Phase 2a.

OTHER OUTCOMES:
Evaluate secondary efficacy measures after 6 months of VRS-317 dosing. | 6 Months
  Secondary efficacy measures during Phase 2a include change in height SDS and change in bone age after 6 months VRS-317 treatment.
Evaluate pharmacodynamic measures | 8 Months
  Secondary outcome measures include evaluation of pharmacodynamics (PD) as measured by IGF-I and IGFBP-3 responses to single dose VRS-317 during Phase 1b and as measured by IGF-I and IGFBP-3 responses to multiple doses of VRS-317 after repeat dosing during Phase 2a. PD measures will be obtained at multiple timepoints during Phase 1b and Phase 2a.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Clovis, California
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Greenwood Village, Colorado
  - Orlando, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Springfield, Massachusetts
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Livingston, New Jersey
  - Morristown, New Jersey
  - Buffalo, New York
  - Mineola, New York
  - Sleepy Hollow, New York
  - Cleveland, Ohio
  - Columbus, Ohio
  - San Antonio, Texas
  - Seattle, Washington